CLINICAL TRIAL: NCT00001999
Title: A Pilot Study to Obtain Preliminary Information Regarding the Efficacy and Safety of the Combination of Immune Globulin and Ganciclovir as Compared to Ganciclovir Alone in the Treatment of Sight-Threatening CMV Retinitis in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American National Red Cross (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 079A; 219-90
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-04

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Gamma-Globulins; Ganciclovir; Drug Therapy, Combination; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Immunization, Passive
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Immunoglobulins; Ganciclovir

INTERVENTIONS:
Drug: Globulin, Immune
Drug: Ganciclovir

SUMMARY:
To evaluate whether immune globulin and ganciclovir (DHPG) results in faster initial response as compared to DHPG alone. To evaluate whether immune globulin and DHPG gives longer duration of remission than DHPG alone (i.e. 16 weeks). To evaluate the toxicities of the combination of DHPG and immune globulin as compared to those of DHPG alone. To evaluate if there is a difference between the two groups in regard to survival, immune functions, and CMV viremia and viruria.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* First episode of sight-threatening CMV retinitis.
* At least one pending culture for CMV from the blood or urine prior to entry.
* Life expectancy > 6 months.
* Karnofsky performance = or > 60.
* Ability to understand the nature of the study, to comply with study requirements, and to sign informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* Known selective IGA deficiency or antibodies against IgA.
* History of previous episodes of sight-threatening CMV retinitis.

Patients with the following are excluded:

* Previous episode of sight-threatening CMV retinitis.
* Concomitant treatment with other investigational agents except ddI or ddC.
* Life expectancy < 6 months.
* Continued alcohol or drug abuse.
* Known selective IgA deficiency and known to have antibodies against IgA.
* Karnofsky performance <60.

Other investigational agents except ddI or ddC.

ddI ddC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown Univ Med Ctr, Washington D.C., District of Columbia, United States